CLINICAL TRIAL: NCT02824211
Title: Demonstrating the Feasibility of a Novel Oxygen Delivery Device in Responding to Real Time Oxygen Needs (The Right Dose System, RDS)
Brief Title: Demonstrating the Feasibility of a Novel Oxygen Delivery Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was unable to obtain funding
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Laren Tan, MD, Assistant Professor of Medicine, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5160199
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Increased Oxygen Demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Right Dose System (Experimental): Use of automated oxygen titration during exertion
  Interventions: Device: Right Dose System

INTERVENTIONS:
Device: Right Dose System — Automated titration of oxygen system during exertion

SUMMARY:
Purpose: To investigate the feasibility of a new oxygen delivery device, the "Right Dose System" (RDS). It delivers individualized boluses of oxygen during rest and exertion to maintain acceptable oxygen saturations.

The procedures include: Enrollment of 10 patients, who are randomized to either exercise with their oxygen prescription followed by exercise with the RDS, or exercise with the RDS followed by exercise on their oxygen prescription. Randomization will occur on a 1:1 basis. Each set of exercise will be separated by a 30 minute recovery session. Subjects will be adults who are on supplemental oxygen and are able to exercise on a treadmill. Subjects will be above 18 years of age. Subject participation will last approximately 1 month. Subjects will be recruited from the Loma Linda pulmonary clinic and the pulmonary rehabilitation program. Consent will take place in the pulmonary clinic, pulmonary function lab or pulmonary rehabilitation by trained study physicians. If Multi-center: N/A (single center) If Single center or investigator-initiated: 10 subjects will participate in the study.

DETAILED DESCRIPTION:
Consent will be administered by trained study physicians-each subject will be given the opportunity to read the IRB approved consent form and ask questions before being enrolled in the study. Consenting investigating physicians are all licensed medical doctors in the state of California and will be instructed to determine that the subject is competent before obtaining consent. After questions and concerns are answered, the patient will sign and date the consent form. This process will be witnessed, signed and dated by one of the clinic staff as well as the investigator.

This is a non-blinded study without a placebo group. The investigators will randomize subject assignment to two cohorts with opposing intervention order.

Subject confidentiality will be maintained by all staff. The LLUH Research Protections HIPPA form will be utilized to inform and gain consent of the subject. Data will be maintained in a locked department, in a locked office and in a locked cabinet. All electronic data will be stored on the LLUH network and servers.

Study Design

Background/Rationale for Study:

The trial is designed to investigate the efficacy and safety of a novel personalized oxygen delivery device called the "Right Dose System" (RDS) compared to standard prescription of oxygen, and current oxygen delivery devices during exercise. As an individual's oxygen needs vary according to their level of activity, RDS would provide an individualized tailored pulse of oxygen to meet the demand of each individual patient while maintaining the appropriate oxygen saturation.

Objectives:

To compare RDS to the standard flow of oxygen on current prescription in patients who require supplemental oxygen during rest and exercise. This is a non-blinded, cross-over study with 1:1 randomization to either intervention A then B, or B then A. It will ascertain the feasibility of this novel oxygen conservation device in maintaining oxygenation saturations during exercise. The goal of the study is to establish proof of concept for this device.

Research Interventions:

During exercise the utilization of the right dose system (RDS) will be compared to patient's standard oxygen therapy. The study subjects will be enrolled to test 2 different oxygen delivery devices (standard oxygen delivery device and RDS with SPO2 measurement).

Visit 1: Screening & Evaluation Patients will be enrolled in clinic or pulmonary rehabilitation. At this time, screening, evaluation and education about the study as well as consent and demographics will be performed at: 1) pulmonary clinic at faculty medical offices (FMO), 2) Loma Linda University Medical Center pulmonary function testing lab and/or 3) Loma Linda University Medical Center pulmonary rehabilitation office.

Visit 2:

Two tests evaluating O2 administration with O2 prescription & RDS with active pulse oximetry separated by a 30 minute recovery period. Order of intervention will be randomized into 2 groups: standard O2 therapy followed by RDS, versus RDS followed by standard O2 therapy.

1. Measuring - exercise time, constant work rate endurance time, SPO2, modified Borg scale for perceived exertion and shortness of breath.
2. The second end point will be how much mean O2 delivered/minute (because patients may be able to exercise much longer on the RDS)

Investigational Device:

* Name of device: Right Dose System
* Manufacturer: Smart Oxygen
* Status with Food & Drug Administration, ID#: Pending Class 2, 5-10K predicate meeting
* Review of animal studies & previous human studies: None
* Reported adverse effects: None, minimal risk device.

Data Collection:

Demographics: Including etiology of hypoxemia, severity of disease process, height, weight, age, gender, oxygen prescription, current oxygen delivery device.

Resting blood pressure Pulse oximetry before, during, and after exercise (using the Masimo Radical 7 pulse oximeter, K120657) Comfort level with walking, Perceived Exertion Level (modified Borg scale) Resting, exercise and post-exercise Shortness of Breath (modified Borg scale) Data Analysis The trial is powered to demonstrate feasibility of RDS in maintaining targeted oxygen saturations in hypoxemic patients with exercise.

Descriptive statistics will be calculated for the baseline variables (demographics, objective, and physical measures)-this will include means, SD, and range. Will evaluate the differences in oxygenation at the three different levels of activity (rest, low exercise, moderate exercise) utilizing the 2 different oxygen delivery systems by repeated measures analysis of variance.

Constant work rate exercise time will be compared between the two groups via paired Student's T-Test.

Will have statistician assistance in providing: 2 variable t-test, ANOVA as will have repeated measures.

Benefits There will be no immediate benefit to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients currently on home supplemental oxygen
* Ambulatory patients able to exercise on treadmill

Exclusion Criteria:

* Prior use of an investigational medicinal product and or investigational medical device within the last month OR planned or concurrent participation in a clinical trial for any investigational drug or investigational device.
* Current Prisoner
* Known to be pregnant
* < 18 years old
* Inability to measure pulse oximetry reliably
* Patients greater than 300 lbs (weight is not supported by our treadmill).
* Patients with known pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Exercise time | Day 2
  Constant work rate testing

SECONDARY OUTCOMES:
Time in targeted oxygen saturation range | Day 2
  Constant work rate testing
Oxygen utilized during exertion | Day 2
  Constant work rate testing

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Nguyen, MD, MS, Study Chair — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No